CLINICAL TRIAL: NCT06122961
Title: Prevalence of Systemic Inflammation in Patients With Atherosclerotic Cardiovascular Disease and Heart Failure
Brief Title: Levels of Inflammation in People With Cardiovascular Disease (POSEIDON)
Acronym: POSEIDON
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN6018-7527; U1111-1286-3420 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Risk; Heart Failure; Chronic Kidney Disease
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Atherosclerotic cardiovascular disease (ASCVD) with chronic kidney disease (CKD): electronic case report form (eGFR) below 60 ml/min/1.73m^2
  Interventions: Other: No treatment given
- ASCVD without CKD: eGFR greater than or equal to 60 ml/min/1.73m^2
  Interventions: Other: No treatment given
- HF with preserved ejection fraction (HFpEF) or HF with mildly reduced ejection fraction (HFmrEF)
  Interventions: Other: No treatment given
- Heart failure (HF) with reduced ejection fraction (HFrEF)
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
This study will collect medical and background information from participants with diseases that affect the heart and blood vessels (cardiovascular disease). Participants will continue their normal care and will not get any treatment other than those the study doctor has prescribed.

ELIGIBILITY:
Inclusion criteria:

1. Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study.
2. Age 18 years or above at the time of signing the informed consent.
3. Presence of ASCVD (atherosclerotic cardiovascular disease) and/or HF (heart failure)
4. Presence of serum creatinine in the medical chart within 24 months prior to signing of informed consent (for ASCVD patients only).

Exclusion criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Current participation (i.e., signed informed consent) in any other interventional clinical study.
3. Any hospitalization or unplanned visit within the last 60 days (including exacerbation of chronic disease with hospitalization).
4. Clinical evidence, or suspicion of, active infection within the last 60 days.
5. Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from cardiology sites reflecting a real-world population of ASCVD and HF patients.
Sampling Method: Non-Probability Sample
Enrollment: 18198 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
High sensitivity C-reactive protein (hsCRP) greater than or equal to 2 mg/L (yes/ no) | At visit (day 0)
  Count of patient

SECONDARY OUTCOMES:
Interleukin 6 (IL-6) | At visit (day 0)
  pg/ml
N-terminal prohormone of brain natriuretic peptide (NT-proBNP) | At visit (day 0)
  pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (195):
- United States (2):
  - Mission Cardiovascular Research Institute, Fremont, California
  - Texas Institute of Cardiology PA, McKinney, Texas
- Argentina (10):
  - Hospital Italiano Regional Sur, Bahía Blanca, Buenos Aires
  - Clínica Coronel Suarez, Coronel Suárez, Buenos Aires
  - Hospital Italiano de la Plata, La Plata, Buenos Aires
  - Centro Médico CIMEL, Lanús Este, Buenos Aires
  - Fundacion Favaloro, CABA, Buenos Aires, Argentina
  - INECO Neurociencias Oroño, Rosario, Santa Fe Province
  - DIM Clinica Privada, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes SRL, Buenos Aires
  - Instituto Médico DAMIC, Córdoba
  - Hospital Luis Lagomaggiore, Mendoza
- Australia (4):
  - Renal Research Gosford, Gosford, New South Wales
  - Advara HeartCare, Auchenflower, Queensland
  - Advara HeartCare, Leabrook, South Australia
  - Barwon Health (The Geelong Hospital), Geelong, Victoria
- Brazil (14):
  - Sociedade Hospitalar Angelina Caron, Brazil, Campina Grande do Sul, Paraná
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - i9 Pesquisas Clínicas, Campinas, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Nucleo de Pesquisa Clinica do Hospital Vera Cruz, Belo Horizonte/MG
  - Hospital do Coração do Brasil, Brasília
  - IPECC - Instituto de Pesquisa Clínica de Campinas, Campinas
  - HC-UFG - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia
  - ICM - Instituto do Coração de Marília, Marília/SP
  - Instituto D'OR de Pesquisa e Ensino, Rio de Janeiro
  - Hospital Ana Nery, Salvador
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, Sao Jose Rio Preto
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo
  - Universidade Federal de Sao Paulo - UNIFESP, São Paulo
- Canada (10):
  - Fraser Clinical Trials Inc., New West Minster, British Columbia
  - North Shore Heart Centre, North Vancouver, British Columbia
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Corcare Cardiovascular Research Inc, Scarborough Village, Ontario
  - Corcare Cardiovascular Research, Scarborough Village, Ontario
  - Winchester Dist Memorial Hosp, Winchester, Ontario
  - [Legal] Viacar Recherches Cliniques, Inc., Brossard, Quebec
  - CardioVasc HR Inc, Saint-Jean-sur-Richelieu, Quebec
  - CIUSSS de la Mauricie-et-du-Centre-du-Québec, Trois-Rivières, Quebec
- China (16):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - NIS-Lanzhou University Second Hospital, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen Universtiy, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - China-Japan Union Hospital of Jilin University-Cardiology, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - The Second Hospital of Shandong University, Jinan
  - The First Affiliated Hospital of Xi'an Jiaotong University-Cardiovascular, Xi'an
- Nemocnice Na Františku, Prague, Czechia
- Denmark (9):
  - Holbæk Sygehus, Holbæk, Region Sjælland
  - Bispebjerg og Frederiksberg Hospital, Frederiksberg
  - Herlev og Gentofte Hospital, Herlev
  - Regionshospitalet Gødstrup, Hjertesygdomme, Herning
  - Hillerød Endokrinologisk amb. H0652, Hillerød
  - Hvidovre Hospital Hjertemedicinsk, Hvidovre
  - Amager Hospital - Medicinsk Amb, København S
  - Rigshospitalet, København Ø
  - Sjællands Universitetshospital_Roskilde, Roskilde
- France (27):
  - Centre Hospitalier Universitaire Amiens Picardie-Site Sud, Amiens
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Saint Andre, Bordeaux
  - Hospices Civils de Lyon-Hopital Cardiologique Louis Pradel-1, Bron
  - Centre Hospitalier Regional Universitaire de Tours-Hopital Trousseau, Chambray-lès-Tours
  - Centre Hospitalier Intercommunal Compiegne - Noyon, Compiègne
  - Centre Hospitalier Universitaire de Dijon-Hopital Le Bocage, Dijon
  - Centre Hospitalier Universitaire Grenoble Alpes-Site Nord Michallon-1, Grenoble
  - Centre Hospitalier de Versailles-Hopital Andre Mignot, Le Chesnay-Rocquencourt
  - Les Hopitaux de Chartres-Hopital Louis Pasteur, Le Coudray
  - Centre Hospitalier Et Universitaire de Limoges-Hopital Dupuytren, Limoges
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Clinique Pont de Chaume, Montauban
  - Centre Hospitalier Universitaire de Montpellier-Hopital Saint-Eloi, Montpellier
  - Centre Hospitalier Universitaire de Nice-Hopital Pasteur, Nice
  - Centre Hospitalier Universitaire de Nimes-Hopital Caremeau, Nîmes
  - Centre Hospitalier Universitaire D'Orleans, Orléans
  - Ap-Hp-Hopital Hotel Dieu Paris, Paris
  - Ap-Hp-Hopital Cochin, Paris
  - Centre Hospitalier de Pau - Hopital Francois Mitterrand, Pau
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Clinique Saint Hilaire, Rouen
  - Centre Hospitalier Universitaire de Nantes-Hopital Nord Laennec-1, Saint-Herblain
  - Aura Paris, Saint-Ouen
  - Centre Hospitalier Intercommunal Toulon La Seine-Sur-Mer - Hopital Sainte Musse, Toulon
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil-1, Toulouse
  - Chru de Nancy - Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (27):
  - Universitätsklinikum Freiburg Herzzentrum, Freiburg im Breisgau, Baden-Wurttemberg
  - SRH Klinikum Karlsbad - Langensteinbach GmbH - Innere Medizin, Karlsbad, Baden-Wurttemberg
  - Med. Universität Lübeck, Lübeck, EK Uni Lübeck
  - Charité - Campus Benjamin Franklin - Klinik für Kardiologie, Angiologie und Intensivmedizin, Berlin
  - Charité - Campus Virchow-Klinikum - Kardiologie, Angiologie und Intensivmedizin (CRU), Berlin
  - Universitätsklinikum Bonn (AöR) - Medizinische Klinik und Poliklinik II - Herzzentrum, Bonn
  - Kardiologisch-Angiologische Praxis Herzzentrum Bremen, Bremen
  - Kath. St. Paulus GmbH - Kardiologie, Dortmund
  - MVZ "Am Felsenkeller" (Dresden), Dresden
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - DaVita Clinical Research Deutschland GmbH, Düsseldorf
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - Universitaetsklinikum Essen - Klinik für Kardiologie und Angiologie, Essen
  - Universitätsklinikum Frankfurt aM - Kardiologie, Frankfurt am Main
  - Klinikum Friedrichshafen GmbH - Klinik für Kardiologie, Angiologie, Pneumologie und internistische Intensivmedizin, Friedrichshafen
  - Universitätsmedizin Göttingen - Dept. Herzzentrum Göttingen, Göttingen
  - UKS - Klinik für Pädiatrische Onkologie und Hämatologie, Homburg/Saar
  - Universitätsklinikum Jena - Kardiologie, Jena
  - Kardiopraxis Schirmer, Kaiserslautern
  - Marienhaus Klinikum Mainz GmbH - Innere Medizin I, Mainz
  - Universitätsmedizin Mainz, Kardiologie I, Studienzentrum, Mainz
  - zero PRAXEN Mannheim-Schwetzingerstadt, Mannheim
  - Klinikum rechts der Isar TU München - Nephrologie, München
  - Universitätsklinikum Tübingen - Innere Medizin III Kardiologie und Angiologie, Tübingen
  - Josephs-Hospital Warendorf - Medizinische Klinik II, Warendorf
  - Al-Zoebi, Wermsdorf
  - Universitatsklinikum Würzburg - Zentrum für Herzinsuffizienz, Würzburg
- India (7):
  - Gauri Heart Centre, Srinagar, Jammu and Kashmir
  - Manoria Heart and Critical Care Hospital, Bhopal, Madhya Pradesh
  - Arneja Heart & Multispeciality Hospital, Nagpur, Maharashtra
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - The Madras Medical Mission, Chennai, Tamil Nadu
  - Shri Mahant Indiresh Hospital, Dehradun, Uttarakhand
  - Apollo Multispeciality Hospital, Kolkata, Kolkata, West Bengal
- Italy (27):
  - Policlinico Mater Domini Università di Catanzaro, Germaneto, Catanzaro
  - Ospedale del Tigullio ASL4 Liguria, Lavagna, Genova
  - Istituto Clinico Humanitas, Rozzano, Milano
  - IRCCS Multimedica, Sesto San Giovanni, Milano
  - IRCCS Policlinico San Donato, San Donato Milanese, Milan
  - Complesso Ospedaliero "Nuovo Ospedale di Rivoli", Rivoli, Torino
  - Ospedale dell'Angelo, Zelarino, Venezia
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - University of Brescia, Brescia
  - AO S. Anna e S. Sebastiano, Caserta
  - Presidio Ospedaliero dell'Annunziata, Cosenza
  - IRCCS Azienda Ospedaliero Universitaria San Martino - IST, Genova
  - Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AORN A. Cardarelli, Napoli
  - Azienda Ospedaliera Universitaria Federico II di Napoli, Napoli
  - A.O.U. Policlinico Giaccone, Palermo
  - Azienda Ospedaliera-Universitaria Parma, Parma
  - AOU Perugia, Perugia
  - Fondazione Toscana G. Monastiero, Pisa
  - ASP Ragusa, Ragusa
  - Arcispedale S Maria Nuova Azienda ULSS-IRCCS, Reggio Emilia
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Fondazione Univ. Policlinico A.Gemelli, Roma
  - AOU Sassari, Sassari
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Azienda Ospedaliera di Udine Ospedale S. Maria della Misericordia, Udine
- Norway (5):
  - Nordland Hospital Trust, Bodø
  - Sykehuset Østfold Kalnes, Grålum
  - Colosseumklinikken Medisinske Senter AS, Oslo
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
  - Skedsmo Medisinske Senter, Norway, Skedsmokorset
- Poland (8):
  - Ind. Prak. Lek. w dziedz. Kardiologii lek. med. K. Cymerman, Gdynia, Pomeranian Voivodeship
  - Specjalistyczna Praktyka Lekarska s.c. Iwona Woźniak Skowerska Mariusz Skowerski, Katowice
  - SPZOZ USK im. Wojskowej Akademii Medycznej UM w Łodzi - Centralny Szpital Weteranów, Lodz
  - Medicome Sp. z o.o., Oświęcim
  - NZOZ Pro-Cordis Sopockie Centrum Bad. Kardiolog., Sopot
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne Sp. z o. o., Szczecin
  - Polsko-Amerykanskie Kliniki Serca.American Heart of Poland Sp. z o.o., Tychy
  - 4 Wojskowy Szpital Kliniczny z Poliklinika SP ZOZ, Wroclaw
- South Korea (19):
  - Gachon University Gil Medical Center, Incheon, Timis
  - Pusan National University Hospital, Busan
  - Daegu Catholic Univ. Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chungbuk National University Hospital, Daejeon
  - Yonsei University Wonju Severance christian hospital, Gangwon-do
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Kyunghee University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Sweden (8):
  - Danderyd sjukhus, Danderyd
  - Medicinkliniken Ryhov, Jönköping
  - Centralsjukhuset Karlstad, Karlstad
  - Skane University Hospital, Lund
  - Universitetssjukhuset Örebro, Örebro
  - Sodersjukhuset AB, Stockholm
  - Karolinska Universitetssjukhuset Solna,FOU Tema Hjärta Kärl, Stockholm
  - Akademiska sjukhuset Uppsala, Uppsala
- Master Centre for United Kingdom, Gatwick, West Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com